CLINICAL TRIAL: NCT03303872
Title: Evaluation of Atrial Fibrillation Occurrence in Sick Sinus and Complete Atrioventricular Block Patients After Pacemaker Implantation (AF-pacemaker Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2017-0008
Record Dates: First submitted 2017-09-17; First posted 2017-10-06 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Post Pacemaker Implantation Patients
Keywords: atrial high rate episode; pacemaker; atrial fibrillation; stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AF-pacemaker registry

SUMMARY:
This study is prospective Cohort study which was performed in multicenter (General Hospital) in Korea. Inclusion criteria is patients post pacemaker implantation. The purpose is to investigate the occurrence of device detected subclinical atrial fibrillation (atrial high rate episode) in patients post pacemaker implantation and assess long term clinical results.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years
* Patients eligible for the indications for permanent pacemaker implantation in accordance with 2016 revised Korean indication guideline on cardiac pacemaker implantation
* Estimated percentage of atrial pacing >40% under sinus rhythm (LR≥60bpm, close hysteresis and rest rate)
* Estimated percentage of ventricular pacing >40% under sinus rhythm (LR≥40bpm, DDD pacing, close hysteresis and rest rate)
* Patients who are willing to sign the informed consent.
* Patients who are willing to receive the implantation and post-operative follow-up.

Exclusion Criteria:

* Persistent or permanent AF
* Severe hepatic and renal insufficiency (AST or ALT ≥ three times of normal upper limit; SCr > 3.5 mg/dl or Ccr < 30ml/min)
* Thyroid gland dysfunction
* Pregnancy
* Malignant tumor
* Severe organic heart disease (such as moderate to severe mitral regurgitation, dilated cardiomyopathy, hypertrophic cardiomyopathy, severe heart valve disease)
* Life expectancy < 12 months
* Patients unable or unwilling to cooperate in the study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients post pacemaker implantation
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-12-31 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of subclinical atrial fibrillation (atrial high rate episode) | 3 months after pacemaker implantation
Occurrence of subclinical atrial fibrillation (atrial high rate episode) | 6 months after pacemaker implantation
Occurrence of subclinical atrial fibrillation (atrial high rate episode) | every 1 year upto 3 years after pacemaker implantation
  Occurrence of subclinical atrial fibrillation (atrial high rate episode) during 36 months (3 years) post pacemaker implant
Occurrence of stroke | 3 months after pacemaker implantation
  Stroke based on device detected subclinical atrial fibrillation episodes
Occurrence of stroke | 6 months after pacemaker implantation
  Stroke based on device detected subclinical atrial fibrillation episodes
Occurrence of stroke | every 1 year upto 3 years after pacemaker implantation
  Stroke based on device detected subclinical atrial fibrillation episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kim M, Kim TH, Yu HT, Choi EK, Park HS, Park J, Lee YS, Kang KW, Shim J, Sung JH, Oh IY, Joung B; AF-Pacemaker Study Group. Prevalence and Predictors of Clinically Relevant Atrial High-Rate Episodes in Patients with Cardiac Implantable Electronic Devices. Korean Circ J. 2021 Mar;51(3):235-247. doi: 10.4070/kcj.2020.0393. PMID 33655723